CLINICAL TRIAL: NCT03074682
Title: Fluid Administration With LifeFlow vs Push/Pull
Brief Title: Novel Device for Rapid Fluid Administration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1612018709
Record Dates: First submitted 2017-02-28; First posted 2017-03-09 (Actual); Results first posted 2019-01-31 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Device Related Sepsis
Keywords: Resuscitation
MeSH Terms: interventions — Double-Balloon Enteroscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Lifeflow (Experimental): Participants in this arm will use the Lifeflow device to administer fluid in a simulation in a simulation setting.
  Interventions: Device: Lifeflow
- Push/Pull (Active Comparator): Participants in this arm will use the Push/Pull method to administer fluid in a simulation in a simulation setting.
  Interventions: Device: Push/Pull
- Pressure Bag (Active Comparator): Participants in this arm will use a Pressure Bag to administer fluid in a simulation in a simulation setting.
  Interventions: Device: Pressure Bag

INTERVENTIONS:
Device: Lifeflow — Following a 5-minute training video where instructions on device are presented to participants, participants are given the device, a 1L NS bag, tubing and a 22g IV. Prior to beginning the simulation, they will demonstrate ability to set up the device and fill an empty container with fluid.
  Arms: Lifeflow
Device: Push/Pull — Following a 5-minute training video where instructions on device are presented to participants, participants are given the device, a 1L NS bag, tubing and a 22g IV. Prior to beginning the simulation, they will demonstrate ability to set up the device and fill an empty container with fluid.
  Arms: Push/Pull
Device: Pressure Bag — Following a 5-minute training video where instructions on device are presented to participants, participants are given the device, a 1L NS bag, tubing and a 22g IV. Prior to beginning the simulation, they will demonstrate ability to set up the device and fill an empty container with fluid.
  Arms: Pressure Bag

SUMMARY:
The aim of the study is to determine if a new device is more effective in fluid administration than devices currently used when resuscitating pediatric patients in septic shock. This study will take place in a simulation lab setting and will not include the use of patients.

DETAILED DESCRIPTION:
In this study, participants will be randomized to one of three devices in a Pediatric Intensive Care Unit simulation setting. Each participant will be provided the device, a 1L NS bag, tubing and a 22g IV. In each scenario, the objective will be to administer 3 20cc/kg boluses within a 15 minute period to the simulated patient.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric emergency medicine or pediatric intensive care unit nurses, pediatric residents, medics and attendings.

Exclusion Criteria:

* Inability to operate equipment due to illness or physical impairment.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-06-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Departments of Pediatrics and Emergency Medicine, Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kline M, Crispino L, Bhatnagar A, Panchal RA, Auerbach M. A Randomized Single-Blinded Simulation-Based Trial of a Novel Method for Fluid Administration to a Septic Infant. Pediatr Emerg Care. 2021 Jun 1;37(6):e313-e318. doi: 10.1097/PEC.0000000000001583. PMID 30106868

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pressure Bag | Push/Pull | Lifeflow
Started | 18 | 18 | 18
Completed | 18 | 18 | 18
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pressure Bag | Push/Pull | Lifeflow | Total
Number analyzed (Participants) | 18 | 18 | 18 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 18 | 18 | 18 | 54
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Gender/sex was not collected for participants.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 18 | 18 | 18 | 54
Provider Type [Count of Participants; unit: Participants]
  MD - Fellow | 2 | 0 | 0 | 2
  MD - Resident | 7 | 8 | 7 | 22
  MD - Attending | 0 | 1 | 2 | 3
  Paramedic | 1 | 1 | 1 | 3
  RN | 8 | 8 | 8 | 24
Patients Cared For [Count of Participants; unit: Participants] — Patients you cared for in the last year requiring rapid volume infusion.
  Participants
    0 | 0 | 1 | 1 | 2
    1-5 | 8 | 8 | 8 | 24
    6-10 | 3 | 3 | 4 | 10
    > 10 | 7 | 6 | 5 | 18
Preferred Method [Count of Participants; unit: Participants] — Preferred method of rapid volume infusion.
  Participants
    Pressure Bag | 7 | 7 | 6 | 20
    Push/Pull | 4 | 7 | 8 | 19
    Rapid Infuser | 2 | 0 | 1 | 3
    Pump/Smart Pump | 4 | 2 | 1 | 7
    Syringe | 0 | 2 | 0 | 2
    MISSING | 1 | 0 | 2 | 3
Simulation Experience [Count of Participants; unit: Participants] — Number of simulation (Sims) trainings per year.
  Participants
    > 5 Sims per Year | 7 | 10 | 9 | 26
    1 -5 Sims per Year | 11 | 8 | 9 | 28
Clinical Team Member Experience [Count of Participants; unit: Participants] — Ever worked clinical with team member?
  Participants
    Yes | 16 | 16 | 16 | 48
    No | 2 | 2 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Successful Administration of 60 mL/kg
Description: Participants will be timed to determine if they are able to administer 60 mL/kg of fluid within a 20 minute timeframe. This outcome will be measured as a dichotomous 'yes' or 'no' as to whether the task was completed successfully. The initial registered primary outcome was changed from 60 cc/kg in 15 minutes to its current format before the study began.
Time Frame: 20 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Pressure Bag | Push/Pull | Lifeflow
Number analyzed (Participants) | 18 | 18 | 18
Participants | 14 | 18 | 16

2. Secondary Outcome: Time to Complete Fluid Administration
Description: Participants will be timed to determine if they are able to administer 60 mL/kg of fluid within a 20 minute timeframe. The time in which they complete the task will be captured in minutes. The initial registered primary outcome was changed from 60 cc/kg in 15 minutes to its current format before the study began.
Time Frame: Up to 20 minutes
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Pressure Bag | Push/Pull | Lifeflow
Number analyzed (Participants) | 18 | 18 | 18
seconds | 718.9 (57.3) | 519.4 (26.3) | 376.5 (30.4)

3. Secondary Outcome: NASA Task Load Index (TLX)
Description: The NASA Task Load Index (TLX) is a series of measures that capture workload. Each scale employs a visual analog scale that measures each of the domains. The domains are Mental Domain, Physical Demand, Temporal Demand, Performance, Effort and Frustration Level. Each scale domain and the Composite has a range from 0 to 100 with 100 being the highest indicator of workload.
Time Frame: 15 minutes
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Pressure Bag | Push/Pull | Lifeflow
Number analyzed (Participants) | 18 | 18 | 18
score on a scale
  Composite | 42.50 [22.08 to 54.79] | 40.42 [22.29 to 48.13] | 30.00 [22.08 to 38.33]
  Mental | 60.00 [43.75 to 75.00] | 57.50 [31.25 to 68.78] | 37.50 [20.00 to 50.00]
  Physical | 20.00 [5.00 to 57.50] | 22.50 [11.25 to 53.75] | 20.00 [5.00 to 50.00]
  Temporal | 55.00 [30.00 to 71.25] | 62.50 [31.25 to 75.00] | 35.00 [23.75 to 51.25]
  Performance | 27.50 [20.00 to 47.50] | 22.50 [10.00 to 37.50] | 25.00 [20.00 to 30.00]
  Effort | 57.50 [30.00 to 75.00] | 50.00 [33.75 to 65.00] | 40.00 [20.00 to 56.25]
  Frustration | 15.00 [5.00 to 40.00] | 17.50 [6.25 to 30.00] | 12.50 [5.00 to 17.50]

4. Other Pre Specified Outcome: Post Intervention Survey
Description: A qualitative questionnaire will be administered to participants following the simulation. Questions include information about experience with various methods and other feedback relevant to evaluation. This outcome was included in the registration is actually captured by the NASA Task Load Index (TLX) that was reported.
Time Frame: 15 minutes
Population: This outcome is analyzed as the NASA Task Load Index (TLX).
Arm/Group | Pressure Bag | Push/Pull | Lifeflow
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Description: This study was conducted using patient simulation and looked at fluid administration across different techniques. The participants in the study were not at risk for adverse events and this information was not collected.
Arm/Group | Pressure Bag | Push/Pull | Lifeflow
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-12-21): https://cdn.clinicaltrials.gov/large-docs/82/NCT03074682/Prot_000.pdf
  • Statistical Analysis Plan (2016-12-21): https://cdn.clinicaltrials.gov/large-docs/82/NCT03074682/SAP_001.pdf